CLINICAL TRIAL: NCT06033196
Title: Targeting Inflammation and Alloimmunity in Lung Transplant Recipients With Tocilizumab (CTOT-45)
Brief Title: Tocilizumab in Lung Transplantation
Acronym: ALL IN LUNG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT CTOT-45
Record Dates: First submitted 2023-08-24; First posted 2023-09-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Transplant
Keywords: Lung Transplant; Tocilizumab; Immunosuppression; ACTEMRA
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tocilizumab Group (Experimental): Subject in this group will receive ACTEMRA(R) (Tocilizumab) ,(six injections over 20 weeks) plus standard triple maintenance immunosuppression of Tacrolimus, Mycophenolate Mofetil, corticosteroids
  Interventions: Drug: Tocilizumab
- Placebo Group (Placebo Comparator): Subject in this group will receive placebo for Tocilizumab (sterile normal saline) plus standard triple maintenance immunosuppression of Tacrolimus, Mycophenolate Mofetil, corticosteroids
  Interventions: Drug: Placebo for Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — The initial dose of tocilizumab will be administered in the operating room before reperfusion of the first lung during the lung transplant surgery.
  6 doses will be given once every four weeks over a 20-week period. The dose is approved for pediatric patients who weigh 30 kg or more
  Other Names: ACTEMRA
  Arms: Tocilizumab Group
Drug: Placebo for Tocilizumab — Placebo 0.9% Sodium Chloride Injection USP (Normal Saline)
  Placebo will be given as a single intravenous dose, volume matched to tocilizumab. Placebo will be administered over a period of approximately 60 minutes; once every four weeks over a 20-week period. The first placebo dose will be during the transplant surgery before reperfusion of the first lung allograft, with 5 subsequent monthly doses
  Arms: Placebo Group

SUMMARY:
This is a trial in which 350 primary lung transplant recipients will be randomized (1:1) to receive either Tocilizumab (six doses over 20 weeks) plus standard triple maintenance immunosuppression or placebo (sterile normal saline) plus standard triple maintenance immunosuppression (Tacrolimus, Mycophenolate Mofetil, corticosteroids).

The primary objective is to test the hypothesis that treatment with triple maintenance immunosuppression plus Tocilizumab (TCZ) is superior to triple maintenance immunosuppression plus placebo (saline) as defined by a composite endpoint of a) CLAD, b) listed for re-transplantation, and c) death

ELIGIBILITY:
Inclusion Criteria:

Study Entry:

1. Subject and/or parent guardian must be able to understand the purpose of the study and willing to participate and sign informed consent/assent
2. Greater than or equal to 30 kg body weight
3. Listed or received for a primary lung transplant
4. No previous or planned desensitization therapy prior to transplant
5. Serum Immunoglobulin G (IgG) level greater than 400 mg/dL. Patients treated with intravenous immune globulin (IVIG) for hypogammaglobulinemia are eligible for enrollment if their serum IgG level is greater than 400 mg/dL 14 or more days after the most recent IVIG treatment
6. For women of child-bearing potential, willingness to use highly-effective contraception; according to the Food and Drug Administration (FDA) Office of Women's Health (http://www.fda.gov/birthcontrol).

   Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used for the duration of the study. Those who choose oral contraception must agree to use a second form of contraception after administration of study drug for a period of 1 year after the last dose of study drug
7. Tested negative for latent TB infection (LTBI) using a PPD or interferon-gamma release assay (i.e., QuantiFERON-TB, T-SPOT.TB) within 1 year prior to transplant or has completed appropriate LTBI therapy within the 1 year prior to transplant
8. Vaccinations must be up to date per the Division of Allergy, Immunology, and Transplantation (DAIT) Guidance for Patients in Transplant Trials

Randomization:

1. Provide written informed consent for the study participation, and agree to continue in the study
2. Received a single or bilateral lung transplant
3. Agreement to use contraception; according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective. Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used for the duration of the study. Those who choose oral contraception must agree to use a second form of contraception after administration of study drug for a period of 1 year after the last dose of study drug
4. Negative physical crossmatch at the time of transplant or a crossmatch result that did not require specific treatment per the site's clinical protocol
5. Underwent bronchoscopy and found to have satisfactory bronchial anastomotic healing
6. No desensitization therapy prior to transplant
7. Negative pregnancy test (serum or urine) for women of child-bearing potential within 48 hours prior to randomization
8. Recipient of lungs that have been supported with ex vivo lung perfusion (EVLP) devices are permitted

Exclusion Criteria:

Study Entry:

1. Listed for multi-organ transplant (e.g., heart-lung, liver-lung, kidney-lung)
2. Prior history of allogeneic organ or cellular transplantation
3. Received treatment to deplete Human Leukocyte Antigens (HLA) antibodies before transplantation
4. Currently breast-feeding a child or plans to become pregnant during the timeframe of the study follow up period
5. History of severe allergic and/or anaphylactic reactions to humanized or murine monoclonal antibodies
6. Known hypersensitivity or previous treatment with ACTEMRA(R) (tocilizumab) within the last 3 months
7. Infection with human immunodeficiency virus (HIV)
8. Hepatitis B virus surface antigen or core antibody positive
9. Hepatitis C virus PCR positive (HCV+) patients who have failed to demonstrate sustained viral remission (2 consecutive PCR or Nucleic Acid Tests (NAT) negative tests at least 24 weeks apart), with or without anti-viral treatment;
10. Chronic infection with Burkholderia cenocepacia or Burkholderia gladioli
11. Non-tuberculous mycobacterial (NTM) pulmonary disease; if there is a history of NTM pulmonary disease, culture conversion is necessary for eligibility
12. Presence of active malignancy or history of malignancy less than 5 years in remission, excluding adequately treated in-situ cervical carcinoma, low grade prostate carcinoma, or adequately treated basal or squamous cell carcinoma of the skin
13. History of hemolytic-uremic syndrome/ thrombotic thrombocytopenia purpura
14. History of demyelinating disorders (e.g., multiple sclerosis, chronic inflammation demyelinating polyneuropathy)
15. Current treatment with alkylating agents such as cyclophosphamide
16. History of gastrointestinal (GI) tract perforation
17. History of inflammatory bowel disease except fully excised ulcerative colitis
18. Any history of diverticulitis (event if not perforated) or confirmed diverticular bleeding. (Diverticulosis is not an exclusion).
19. Patients with a platelet count < 100,000/mm^3 (last measurement within 7 days prior to enrollment)
20. Patients with an absolute neutrophil count (ANC) < 2,000/mm^3 (last measurement within 7 days prior to enrollment)
21. Patients with Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) levels >3 times upper limit of normal
22. Patients who use illegal drugs
23. Smoking or vaping within 6 months of listing for transplant
24. Use of investigational drugs within 4 weeks prior to enrollment
25. Any condition that in the opinion of the site Principal Investigator (PI) introduces undue risk by participating in this study

Randomization:

1. Recipient of multi-organ or tissue transplants
2. Clinically stable, without clinical evidence of untreated infection
3. Received a live virus vaccine within 30 days prior to randomization
4. Received treatment to deplete HLA antibodies before transplantation to improve the possibility of transplantation
5. Patients with known donor-specific antibody that will require intervention based on local clinical protocols
6. History of GI tract perforation
7. History of inflammatory bowel disease except fully excised ulcerative colitis
8. History of diverticulitis (diverticulosis is not an exclusion) or diverticular bleeding
9. History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies
10. Known hypersensitivity to ACTEMRA® (tocilizumab)
11. Previous treatment with ACTEMRA® (tocilizumab) within the last 3 months.
12. Recipient or donor with infection with human immunodeficiency virus (HIV)
13. Recipient with hepatitis B virus surface antigen or hepatitis B core antibody positive
14. Hepatitis B negative transplant recipient that received a transplant from a Hepatitis B core antibody positive donor unless the recipient has a Hepatitis B Surface Antigen (HBsAb) titer >10U/L
15. Recipient of a hepatitis C virus nucleic acid test (NAT) positive donor organ
16. Latent TB infection (LTBI) and has not completed appropriate therapy
17. Chronic infection with Burkholderia cenocepacia or Burkholderia gladioli
18. Non-tuberculous mycobacterial (NTM) pulmonary disease; if there is a history of NTM pulmonary disease, culture conversion is necessary for eligibility
19. Presence of active malignancy (except for non-melanoma skin cancer)
20. History of hemolytic-uremic syndrome/ thrombotic thrombocytopenia purpura
21. History of demyelinating disorders (e.g., multiple sclerosis, chronic inflammation demyelinating polyneuropathy)
22. Current treatment with alkylating agents such as cyclophosphamide
23. Patients with AST or ALT levels > 1.5 times upper limit of normal (last measurement within 1 day prior to randomization)
24. Patients with platelet count <100,000/mm^3 (last measurement within 1 day prior to randomization)
25. Patients with an absolute neutrophil count (ANC) <2,000/mm^3 (last measurement within 1 day prior to randomization)
26. Patients who are administered anti-thymocyte globulin as induction therapy in the immediate post- transplant period
27. Patients who have been treated in the past 3 months, or for whom it is anticipated that treatment with any immunomodulatory biological agents post-transplant are excluded
28. Use of an investigational drug after transplant
29. Smoking or vaping since enrollment
30. Any condition that in the opinion of the site PI introduces undue risk by participating in this study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who meet any one of the pre-specified events detailed in the outcome description: from Baseline up to 36 months | Over a period of 3 years after randomization
  1. The development of Chronic Lung Allograft Dysfunction (CLAD)
     * The development of any form of CLAD will be defined according to the standard 2019 The International Society for Heart and Lung Transplantation (ISHLT) criteria.
  2. Listed for re-transplantation
     * Re-transplantation defined as the subject has been formally registered on the United Network for Organ Sharing (UNOS) waiting list to undergo a second lung transplant surgery
  3. Death
     * Primary analysis will be conducted according to an Intent-to-treat (ITT) principle and therefore will include all randomized subjects who receive Tocilizumab(TCZ) or placebo. The time from randomization to development of CLAD will be compared between the two treatment groups (TCZ vs. placebo) using a Pearson's chi-square test.

SECONDARY OUTCOMES:
Time to the onset of CLAD, being listed for re-transplantation, or death | At 3 years after randomization
Cumulative incidence of Chronic Lung Allograft Dysfunction (CLAD) | At 3 years after randomization
Cumulative incidence listed for re-transplantation | At 3 years after randomization
Cumulative incidence of death | At 3 years after randomization
Freedom from Acute Cellular Rejection (ACR) grade >=A2 | At 3 years after randomization
  Transbronchial lung biopsies will be performed according to the local center standard of care using the 2007 International Society for Heart and Lung Transplantation (ISHLT) criteria.
  Acute Cellular Rejection (A grade Rejection) Scale:
  * None (A0)
  * Minimal (A1)
  * Mild (A2)
  * Moderate (A3)
  * Severe (A4)
  * Ungradable (AX)
Proportion of subjects free from Antibody Mediated Rejection (AMR) | At 3 years after randomization
  Antibody mediated rejection studies will be performed using original H&E stained slides, trichrome/elastic trichrome stain, and C4d immunostain (5 slides per case), along with positive controls
Proportion of subjects free from the development of de novo donor specific antibodies (dnDSA) | At 3 years after randomization
Incidence of Gastrointestinal (GI) tract perforation | At 3 years after randomization
Incidence of serious infections requiring intravenous antimicrobial therapy and need for hospitalization | At 3 years after randomization
Incidence of confirmed bacterial infection requiring antimicrobial therapy | At 3 years after randomization
Incidence of confirmed Cytomegalovirus (CMV) infection requiring antimicrobial therapy | At 3 years after randomization
Incidence of confirmed mold infection requiring antimicrobial therapy | At 3 years after randomization
Incidence of confirmed mycobacterial infection requiring antimicrobial therapy | At 3 years after randomization
Incidence of confirmed community-acquired respiratory viral infection, including coronavirus disease 2019 (COVID-19) infection | At 3 years after randomization
Incidence of discontinuation of Tocilizumab (TCZ) due to an adverse event | At 3 years after randomization
Incidence of discontinuation of Tocilizumab (TCZ) due to serious adverse event | At 3 years after randomization
Incidence of discontinuation of Tocilizumab (TCZ) placebo due to an adverse event | At 3 years after randomization
Incidence of discontinuation of Tocilizumab (TCZ) placebo due to serious adverse event | At 3 years after randomization
Incidence of malignancy excluding squamous or basal cell skin cancer | At 3 years after randomization
Incidence of Tuberculosis (TB) | At 3 years after randomization
Incidence of Post-transplant lymphoproliferative disorder (PTLD) | At 3 years after randomization
Time to the onset of Chronic Lung Allograft Dysfunction (CLAD) | At 3 years after randomization
Time to the onset of being listed for re-transplantation | At 3 years after randomization
Time to the onset of death | At 3 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Joren Madsen, MD, D.Phil., Principal Investigator — Massachusetts General Hospital; Ramsey Hachem, MD, Study Chair — University of Utah Medical Center; Daniel Kreisel, M.D., Study Chair — Washington University School of Medicine
Locations (20):
- United States (20):
  - St. Joseph's Hospital and Medical Center (Site #: 71192), Phoenix, Arizona
  - Cedars Sinai Medical Center (Site #: 71146), Los Angeles, California
  - David Geffen School of Medicine at UCLA (Site #: 71123), Los Angeles, California
  - University of Florida Shands Hospital (Site #: 71131), Gainesville, Florida
  - Emory University (Site #: 71103), Atlanta, Georgia
  - University of Maryland Medical Center (Site #: 71138), Baltimore, Maryland
  - Massachusetts General Hospital (Site #: 71107), Boston, Massachusetts
  - Boston Children's Hospital and Harvard Medical School (Site #: 71001), Boston, Massachusetts
  - Mayo Clinic Rochester (Site #: 71160), Rochester, Minnesota
  - Barnes Jewish Hospital/ Washington University SOM (Site #: 71191), St Louis, Missouri
  - St. Louis Children's Hospital of Washington University (Site #: 71006), St Louis, Missouri
  - Columbia University Medical Center (Site #: 71113), New York, New York
  - Duke University Medical Center (Site #: 71139), Durham, North Carolina
  - Cleveland Clinic (Site #: 71101), Cleveland, Ohio
  - Ohio State University Medical Center (Site #: 71196), Columbus, Ohio
  - Temple University (Site #: 71197), Philadelphia, Pennsylvania
  - University of Texas Southwestern (Site #: 71187), Dallas, Texas
  - Houston Methodist Hospital (Site #: 71120), Houston, Texas
  - University of Texas Health Science at San Antonio (Site #: 71198), San Antonio, Texas
  - University of Utah Medical Center (Site #: 71126), Salt Lake City, Utah

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: NIAID Transplant Programs website — http://www.niaidtransplantstudies.org/